CLINICAL TRIAL: NCT06379139
Title: Dynamic Full-field Optical Coherence Tomography for Endotracheal Tube Biofilm Characterization in Critically Ill Patients
Brief Title: Dynamic Full-field Optical Coherence Tomography for Structural and Microbiological Characterization of Endotracheal Tube Biofilm in Critically Ill Patients
Acronym: BIOPAVIR2
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: MALDINEY J'InvEst-I 2022
Record Dates: First submitted 2024-04-04; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Healthcare Associated Infection; Critically Ill; Endotracheal Tube
MeSH Terms: conditions — Cross Infection; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BIOPAVIR 2 cohort: Adult critically ill patients (> 18 years of age) exposed to endotracheal tube for at least two calendar days
  Interventions: Other: •Dynamic Full-Field Optical Coherence Tomography analysis of endotracheal tube

INTERVENTIONS:
Other: •Dynamic Full-Field Optical Coherence Tomography analysis of endotracheal tube — Dynamic full-field optical coherence tomography analysis of endotracheal tube sections to better apprehend strucural characterization of endotracheal tube-deposited biofilm

SUMMARY:
Biofilm is a microstructure organised into aggregates of microbiological species within a polymeric matrix. As early as the 2000s, the Centers for Disease Control and Prevention (CDC) recognised the possible role of the biofilm lining endotracheal endotracheal tubes in the development of ventilator-associated pneumonia (VAP) , the most common infection in intensive care, with a high morbidity and mortality rate and a significant increase in hospital costs.

Targeting biofilm therefore now appears to be a new area of interest for limiting the risk of VAP, and this rationale has led to the development of an intraluminal for abrading biofilm deposited on the inside of the intubation probe

. Evaluation of this type of strategy nevertheless justifies the introduction of more precise methods for characterisation of the biofilm.

To this end, the investigator carried out an initial clinical study describing the biofilm on intubation probes, BIOPAVIR 1, showing the existence of several biofilm structures, each associated with a specific microbiological signature. Several limitations including a lack of power due to an insufficient number of patients and the use of number of patients, and the use of a confocal microscopy technique with poor axial without the possibility of acquiring metabolic images of the biofilm.

Based on the previous description of biofilm by optical coherence tomography (OCT), and a recent experience with an optimised form of high-resolution OCT, called full-field OCT, the investigator hypothesise that full-field OCT will allow more accurate characterisation of biofilm, due to its high spatial resolution and its potential ability to capture metabolic activity in the biofilm BIOPAVIR 2 proposes to use the performance of full-field OCT to better characterise the biofilm lining endotracheal tubes in patients undergoing mechanical ventilation in intensive care units. This project represents a first step towards understanding the link between the development of biofilm on intubation and the occurrence of VAP

ELIGIBILITY:
Inclusion Criteria:

* Patient or relative informed of the study and having declared their nonobjection
* Patient over 18 years of age
* Patient exposed to mechanical ventilation for at least two calendar days

Exclusion Criteria:

* Patient unable to declare their nonobjection
* Patient whose endotracheal tube collection is impossible
* Patient whose endotracheal tube is collected following self-extubation (sample contamination)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient over 18 years of age having declared their nonobjection and exposed to mechanical ventilation for at least two calendar days
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Dynamic Full-Field Optical Coherence Tomography-based biofilm structure type | At Day 0, within 72hours following endothracheal tube removal
  shape data
type of microbiological associated with each shape | At Day 0, within 72hours following endothracheal tube removal

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MALDINEY, Principal Investigator — CH William Morey
Locations (2):
- France (2):
  - CH William Morey, Chalon-sur-Saône
  - CHU Dijon Bourgogne, Dijon